CLINICAL TRIAL: NCT01507298
Title: An Observational Study to Compare the Outcomes of Ambulatory Gastrointestinal Investigations With Physical Activity Using Accelerometry.
Brief Title: Physical Activity and Gastrointestinal Investigations
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: CRO1766
Record Dates: First submitted 2012-01-06; First posted 2012-01-10 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-08

CONDITIONS: Gastro-oesophageal Reflux Disease
Keywords: Physical activity; Accelerometry; Oesophageal pH; Capsule endoscopy
MeSH Terms: conditions — Gastroesophageal Reflux; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Capsule endoscopy
- 24 hour oesophageal pH study

SUMMARY:
This is an observational study, which aims to compare the outcomes of ambulatory gastrointestinal investigations with physical activity using accelerometry. An ambulatory study refers to one in which the patient is monitored freely, often outside of the hospital environment. For this the investigators will use a lightweight (7.4g) tri-axial accelerometer worn behind the ear.

Hypothesis 1 There is no change in the amount or nature of physical activity taken by patients during ambulatory oesophageal pH monitoring or capsule endoscopy.

Hypothesis 2 There is no correlation between physical activity levels and speed of gastrointestinal transit.

DETAILED DESCRIPTION:
For capsule endoscopy, the investigators are interested in how physical activity affects the speed of capsule transit through the GI tract. Capsule endoscopy involves a patient swallowing a pill which contains a camera, in order to image the parts of the bowel that a conventional endoscope cannot reach. A rapid transit may result in insufficient mucosal visualisation, which would reduce the sensitivity of the investigation.

For oesophageal pH monitoring, it is essential that the patient behaves as they would normally to produce measurements that represent a standard day. Using accelerometry, the investigators can compare the amount, and nature, of physical activity taken throughout the investigation to that of the preceding day, or week. In addition, further analysis of motion data captured will allow us to correlate specific activities and body orientation with pH readings to get a better insight into the pathophysiology of a patient's condition.

The studies will be conducted over 6-9 months in Imperial College Trust's medical outpatient service. All patients undergoing capsule endoscopy or ambulatory oesophageal monitoring will be asked to consider participating. Patients will receive the eAR sensor up to 2 days before their investigation, and will be asked to wear it until the end of their investigation (not whilst sleeping). Capsule endoscopy normally takes less than 12 hours, and pH monitoring takes between 24 and 48 hours. Participation makes no difference to the standard or type of care that they will receive, the sensor data is additional.

ELIGIBILITY:
Inclusion Criteria:

* Planned 24 hour oesophageal pH monitoring study, or capsule endoscopy

Exclusion Criteria:

1. Undergone previous capsule endoscopy or ambulatory oesophageal pH test
2. Currently a hospital in-patient
3. Severe mobility disorder (unable to walk or mobilise independently)
4. Age less than 18 or above 65
5. Physically unable to wear eAR sensor (eg. bilateral hearing aids or particularly small ears)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those who have been advised to undergo 24 hour oesophageal pH monitoring, or capsule endoscopy (from GI outpatients clinic)
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Kwasnicki, BSc Hons, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kwasnicki RM, Ley Greaves R, Ali R, Gummett PA, Yang GZ, Darzi A, Hoare J. Implementation of objective activity monitoring to supplement the interpretation of ambulatory esophageal PH investigations. Dis Esophagus. 2016 Apr;29(3):255-61. doi: 10.1111/dote.12312. Epub 2015 Jan 27. PMID 25625191
- See also: Link to paper showing results of study — http://www.ncbi.nlm.nih.gov/pubmed/25625191

RESULTS

PARTICIPANT FLOW:
Groups:
- Capsule Endoscopy: A pill camera used for imaging the small bowel
- 24 Hour Oesophageal pH Study: Patients wore the accelerometer before and during the ambulatory oesophageal pH test for activity levels to be recorded and compared.
Period: Overall Study
Arm/Group | Capsule Endoscopy | 24 Hour Oesophageal pH Study
Started | 1 | 20
Completed | 1 | 14
Not Completed | 0 | 6
Not completed — Protocol Violation | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Capsule Endoscopy | 24 Hour Oesophageal pH Study | Total
Number analyzed (Participants) | 1 | 20 | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35 (0) | 53 (11) | 50 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 10 | 10
  Male | 1 | 10 | 11
Region of Enrollment [Number; unit: participants]
  United Kingdom | 1 | 20 | 21

OUTCOME MEASURES:

1. Primary Outcome: Physical Activity Change (%)
Description: The primary outcome measure is amount of physical activity undertaken by participants throughout the study period. Participant motion data will be collected using a tri-axial accelerometer in the eAR sensor. Signal processing methods will be used to produce an activity index in the form of a numerical value, from the raw data.
  Activity levels were grouped at 1- minute intervals into restful, low, moderate or high intensity activity.
  Activity levels were calibrated for each participant, classifying activity into quartiles, where the most inactivity was labelled 'Restful', 2nd quartile 'low intensity', 3rd quartile 'moderate intensity' and upper quartile 'high intensity'. This provided a personalised activity profile with which to compare activity during the investigation.
Time Frame: Difference between baseline (2 days average) and test day (during pH monitoring)
Population: Due to significant differences in expected and actual recruitment for the capsule endoscopy arm (i.e. 1 subject), raw data collected were not analysed to produce activity metrics.
Measure: Mean (Standard Deviation); unit: Percentage change in activity
Arm/Group | Capsule Endoscopy | 24 Hour Oesophageal pH Study
Number analyzed (Participants) | 0 | 13
Percentage change in activity |  | -22 (20)

2. Secondary Outcome: Change in Relative Intensity of Daily Activities (%)
Description: Measuring the changes in restful (activity equivalent to sitting), low (activity equivalent to a slow walk), moderate (activity equivalent to a brisk walk) and high intensity activity (activity equivalent to running).
  Including subject-specific activity intensity quartiles, were calculated and compared.
Time Frame: Difference between baseline (2 days average) and test day (during pH monitoring)
Population: Raw data captured for capsule endoscopy group not analysed to produce activity metrics due to insufficient numbers recruited (i.e. 1 subject).
Measure: Mean (Standard Deviation); unit: Percentage change in activity
Arm/Group | Capsule Endoscopy | 24 Hour Oesophageal pH Study
Number analyzed (Participants) | 0 | 13
Percentage change in activity
  Restful |  | 8.5 (17)
  Low |  | -1 (24)
  Moderate |  | -1 (24)
  High |  | -6 (7)

ADVERSE EVENTS:
Time Frame: 2 days
Description: No adverse events were anticipated from participation in this study.
Groups:
- Capsule Endoscopy: A pill camera used to image the small bowel.
Arm/Group | Capsule Endoscopy | 24 Hour Oesophageal pH Study
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/20
Other Adverse Events (participants affected / at risk) | 0/1 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes